CLINICAL TRIAL: NCT05574049
Title: Weight Loss and Therapeutic Metablic Effects of Tetrahydrocannabivarin (THCV) Impregnated Mucoadhesive Strips
Brief Title: Weight Loss, Blood Sugar and Blood Lipid Effects of Tetrahydrocannabivarin (THCV) Impregnated Mucoadhesive Strips
Acronym: THCV
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical Life Care Planners, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Weight Loss with THCV
Record Dates: First submitted 2022-10-03; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Metabolic Syndrome; Morbid Obesity; Hypercholesterolemia; Hyperglycemia
Keywords: tetrahydrocannabivarin; cannabidiol; metabolic syndrome; endocannabinoid system; cannabinoid one receptor
MeSH Terms: conditions — Metabolic Syndrome; Obesity, Morbid; Hypercholesterolemia; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Subjects will be divided into three groups for daily doses. One group with get single dose (8mg THCV/10mg CBD), one group will get double dose (16mg THCV/20mg CBD) and the placebo group will get mouth strip only.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The physician investigator, and all of the test subjects will be masked from knowing which intervention that they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single Dose (Active Comparator): Once daily mouth strip containing 8mg of THCV and 10mg of CBD
  Interventions: Drug: Tetrahydrocannabivarin; Other: Placebo
- Double Dose (Active Comparator): Once daily mouth strip containing 16mg of THCV and 20mg of CBD
  Interventions: Drug: Tetrahydrocannabivarin; Other: Placebo
- Placebo (Placebo Comparator): Once daily mouth strip containing nothing
  Interventions: Drug: Tetrahydrocannabivarin

INTERVENTIONS:
Drug: Tetrahydrocannabivarin — The subjects will take once daily oromucosal strip with intervention drug for 90 days.
  Other Names: THCV
Other: Placebo — The subjects will take once daily oromucosal strip with no drug on it for 90 days
  Other Names: Plain mucoadhesive mouth strip
  Arms: Double Dose; Single Dose

SUMMARY:
The goal of this clinical trial is to compare the efficacy of two different daily doses of tetrahydrocannabivarin impregnated mouth strips in healthy non-diabetic obese adults. The main questions to answer are:

* Is the low dose treatment superior to placebo for losing weight, abdominal girth, cholesterol levels and blood glucose levels?
* Is the low dose treatment superior to placebo for losing weight, abdominal girth, cholesterol levels and blood glucose levels?
* Is one dose better than the other dose?

Participants will take either the low dose, high dose or placebo dose daily for ninety days and have physical measurements and blood tests obtained at the beginning and the end of the study.

DETAILED DESCRIPTION:
Fifty-six adults who met the clinical criteria for obesity (BMI ≥ 30) without comorbid diabetes or cardiovascular disease will be selected for this study. Social media outreach and advertising will be used to identify potential subjects. Prior to starting the study, all subjects will undergo an entrance examination by a blinded independent physician to confirm that they did not have diabetes, active cardiovascular disease, or other confounding health conditions. Initial and final biometric measurements will be taken to include blood pressure, blood oxygen, temperature, height, weight, and abdominal girth. Due to the natural fluctuations in weight, abdominal girth and blood pressure that tend to occur throughout the menstrual cycle, those study participants with active menstrual periods will be scheduled to have their ending biometrics taken during the same phase of their menstrual cycle as when they had their initial biometrics taken, approximately 90 days later. Fasting bloodwork will include a lipid profile, blood sugar, HgbA1c, liver and kidney function studies. LabCorp Inc. will be used for all blood testing.

Each subject will assigned at random to one of three groups: Group A (single dose group), Group B (double dose group,) and Group P (placebo/control group). Subjects will be provided with a 90-day supply of their respective dose (based on group assignment), and instructed to take their assigned dose by mouth, once per day in the morning on an empty stomach. All subjects will be asked to agreed from the outset to refrain from the use of cannabis, CBD, or other hemp-related products throughout the duration of the study. Subjects will be advised to make no changes in their diet or exercise routines.

Each subject will be sent a daily reminder via text message when it was time to take their dose, and was asked to reply with confirmation once they had taken their dose. Additionally, they will be invited to provide feedback on any adverse effects or questions.

ELIGIBILITY:
Inclusion Criteria:

Adults who met the clinical criteria for obesity (BMI ≥ 30) without comorbid diabetes or cardiovascular disease were selected for this study.

Exclusion Criteria:

Under age 18 BMI less than 30 presence of diabetes or cardiovascular disease.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 90 days
  Change in body weight measured in kilograms
Decreased abdominal girth | 90 days
  Change in abdominal girth measures in centimeters
Systolic and diastolic blood pressure | 90 days
  Changes in systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Aspartate Aminotransferase (AST) changes | 90 days
  Change in AST level in blood tests
Alanine Transaminase (ALT) changes | 90 days
  Change in ALT level in blood tests

CONTACTS AND LOCATIONS:
Locations (1):
- Hair and Scalp Clinic, Clearwater, Florida, United States